CLINICAL TRIAL: NCT03913390
Title: Descriptive Study on Decision Making With a Bioethical Perspective in Some Cities of Mexico
Brief Title: Decision Making With Bioethical Perspective in Palliative Care en Mexico
Status: Completed | Type: Observational
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Rosa Margarita Alvarez Alvarez, Principal investigator, University of Guadalajara
Other Study IDs: 218901374
Record Dates: First submitted 2019-04-07; First posted 2019-04-12 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Palliative Care
Keywords: Guideline; Decision Making; Bioethics; Palliative Care; Terminal Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
All clinical practice includes decision making, and sometimes you are ethically challenging because of the consequences it will bring to the patient, the health professional or society in general. Ethics seeks the best solution to a better treatment and seeks to increase the quality of life of the patient with correct decision making. Ethical / bioethical considerations are of a generic nature, and do not apply to specific situations. Therefore, it is suggested that there should be guidelines or recommendations in the field of palliative care in Mexico that may be an adjunct to decision making. The relevance of knowledge, application and management of ethical / bioethical recommendations is unknown as part of decision-making by professionals dedicated to palliative care in our country, taking into consideration the principles of autonomy, beneficence, non-malfeasance and Justice. It is necessary to consider the participation of patients, caregivers and health personnel in this decision making process of decisions. This study intends to identify the current situation of this issue in Mexico.

To analyze the characteristics of decision-making with bioethical involvement in palliative care in a representative sample of care professionals in some regions of the country.

Quantitative method:

* Describe the current situation in decision-making with bioethical involvement in palliative care.
* Identify if the personnel dedicated to palliative care know guidelines or recommendations related to decision-making in palliative care and the current legal framework.
* Know the strategies that palliative care personnel follow in situations in which the decision to make is difficult or problematic.

Qualitative method:

* Know the particular situations that signify a conflict or situation with bioethical implications for health professionals in palliative care.
* Analyze the variables that influence decision-making around the application of bioethics in palliative care.

DETAILED DESCRIPTION:
Mixed study, for the quantitative part, it was prospective, descriptive, and cross-sectional investigation; on the qualitative part it was a case study. A sample of 72 health professionals was considered for the quantitative part and 8 for the qualitative part. The sampling strategy was for convenience. Data collection was achieved through a semi-structured survey applied in a virtual environment with the Google Forms platform. The quantitative data analysis was with descriptive measures of central tendency using the Statistical Package for the Social Sciences 21® (SPSS) software, and the qualitative ones with thematic content analysis techinique through the Qualitative Data Analysis Atlas Ti version 6.0® software.

Informed consent was obtained from the participants for the use of the data.

ELIGIBILITY:
Inclusion criteria for the quantitative sample:

* Agree to participate in the study.
* Health personnel engaged in palliative care
* Work in the public and/or private sector.

Non- inclusion criteria:

* Incomplete survey.

Elegibility criteria for the qualitative sample:

* The participants who answered questions 19 and 20 of the survey sent by Google Forms were chosen.
* Of these, the profession of origin was identified to select those that belonged to professions that are from the disciplines that make up the multidisciplinary teams in palliative care, additionally; The time of work experience in this area was considered, they were included with more than 10 years of experience and less than 10.
* Likewise, the variability of cases and those that reflected an ethical conflict were looked for.

Ineligibility criteria for the qualitative sample:

* Those cases where similar situations or scenarios were described were discarded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Quantitative sampling:
  Non-probabilistic sampling for convenience, of an open nature. Aimed at a specific professional profile according to the theme, the study identified the characteristics of decision-making of the health personnel working in the context of palliative care in different cities of Mexico, the result was not considered generalizable. The Statistical Package for the Social Sciences 21® (SPSS) software was used for statistical analysis.
  Qualitative sampling:
  A sampling called critical case was followed, according to which cases are chosen based on characteristics that can provide different perspectives on the phenomenon, this choice was based on the profession of the participant, the years of seniority in palliative care and that the cases reflected a bioethical conflict or dilemma. Qualitative Data Analysis Atlas Ti version 6.0® software was used for statistical analysis.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Quantitative results | 1 year
  Demographic data, Bioethics training, Experience with clinical situations with bioethical implication.
Qualitative results | 1 year
  The last two questions with a qualitative approach, the objective is to obtain a broader view of the characteristics of decision-making, considering that palliative care by definition is an approach to care from different disciplines

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Ramos-Zuñiga, MD PhD, Study Director — University of Guadalajara
Locations (1):
- Rosa Margarita Alvarez Alvarez, Zapopan, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Undecided